CLINICAL TRIAL: NCT06512389
Title: Evaluating Cannabidiol as a Novel Anticraving Medication for Alcohol Use Disorder: A Human Laboratory Study
Brief Title: Evaluating Cannabidiol as a Novel Anticraving Medication for Alcohol Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021/102
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; cannabidiol; alcohol consumption; craving
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Solutions

STUDY DESIGN:
Intervention Model Description: Within-subject randomized double-blind placebo controlled crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol (Experimental): 10-day supply of 600 mg of CBD, taken orally twice daily
  Interventions: Drug: Oral solution
- Placebo (Placebo Comparator): 10-day supply of 600 mg of placebo, taken orally twice daily
  Interventions: Drug: Oral solution

INTERVENTIONS:
Drug: Oral solution — 300 mg taken morning and evening

SUMMARY:
This human laboratory study aims to assess the effects of cannabidiol on alcohol consumption and craving in participants with alcohol use disorder. In this double-blind within-subject placebo-controlled crossover trial, participants will be randomized to receive both cannabidiol and placebo with a 2-week washout period separating the two treatment phases.

DETAILED DESCRIPTION:
Participants with alcohol use disorder will receive treatment daily (600mg cannabidiol or placebo), each for 10 consecutive days, with a 2-week long washout period between treatments. Participants will be randomized to receive placebo or cannabidiol first (in blocks of random size) so that equal number of participants are allocated to each sequence. Around day 8 of each treatment period, participants will complete an alcohol self-administration session in the laboratory to assess the effects of treatment on alcohol consumption and alcohol-related craving.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-5 criteria for AUD.
* Meets drinking criteria of average weekly consumption > 10 standard drinks for women and > 15 standard drinks for men over the past 90 days.
* Willing to take study medication and participate in laboratory sessions requiring self-administration of alcohol
* Agrees not to use cannabis or illicit drugs during the study period.
* Able to communicate and provide informed consent in English.
* Alanine Aminotransferase (ALT) and Aspartate Transaminase (AST) level should not be more than 2 times the upper normal limit, and bilirubin should not be more than 1.5 times the upper normal limit.
* Enrolled in the Ontario Health Insurance Plan (OHIP)
* Willing and able to safely abstain from alcohol for at least 12 hours prior to the eligibility and alcohol self-administration visit.
* Individuals who are capable of becoming pregnant: agree to the use of highly effective contraception during study participation and for an additional 28 days after the end of cannabidiol administration.

Exclusion Criteria:

* Clinical Institute Withdrawal Assessment (CIWA-Ar) score of 10 or above upon initial assessment
* History of severe alcohol withdrawal including withdrawal seizures, alcoholic hallucinosis, or delirium tremens
* Any history of seizures
* Serious unstable medical condition, including severe hepatic abnormalities
* Having any clinical condition, drug sensitivity, or prior therapy which, in the investigator's opinion, makes the participant unsuitable for the study
* Current medical conditions, prescriptions, or over the counter medications that interfere with receiving the study drug or alcohol (based on the study physician's assessment)
* Severe mental illness (e.g. active psychosis with ongoing delusions and/or hallucinations, active manic or hypomanic episodes, evidence of a major neurocognitive disorder, etc.) and other substance use disorders (moderate or severe; excluding tobacco use disorder) as determined by the qualified investigator
* Experiencing active suicidal ideation within the past 1 month and/or suicide attempt within the past 6 months
* Recent recreational drug use (assessed via urine toxicology screen) other than alcohol and nicotine products
* Current use of CBD products or use of CBD products within the past month.
* History of hypersensitivity to CBD
* Self-report of significant alcohol-induced flushing after 1-2 drinks (a proxy for aldehyde dehydrogenase deficiency)
* Currently pregnant or breastfeeding or intending to become pregnant or breastfeed.
* Currently institutionalized which refers to a person who lives in an institutional collective dwelling, such as a hospital, nursing home or prison, including a resident under custody (e.g., patient or inmate).
* Currently in treatment for AUD (e.g. Alcoholics Anonymous, group therapy, individual therapy, on anticraving medication)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total number of drinks administered during the alcohol-self administration session | 2 hours
  Number of drinks consumed during the alcohol self-administration session.
Peak breath alcohol concentration during the alcohol-self administration session | 2 hours
  Maximum breath alcohol concentration during the alcohol self-administration session.
Craving at baseline as measured by the Alcohol Urge Questionnaire during the alcohol self-administration session. | Baseline
  Alcohol Urge Questionnaire Scores (minimum score = 8; maximum score = 56; higher scores indicates higher levels of craving)
Craving following the priming dose of alcohol as measured by the Alcohol Urge Questionnaire during the alcohol self-administration session. | 20 min after priming dose
  Alcohol Urge Questionnaire Scores (minimum score = 8; maximum score = 56; higher scores indicates higher levels of craving)

SECONDARY OUTCOMES:
Subjective effects of alcohol during the alcohol self-administration session as measured by the Drug Effects Questionnaire. | 3 hours
  Drug Effects Questionnaire (each item scored from 0 to 100). The higher the score, the more the participant feels that "effect".
Subjective effects of alcohol during the alcohol self-administration session as measured by the Brief Biphasic Alcohol Effects Scale | 3 hours
  Brief Biphasic Alcohol Effects Scale (stimulation factor ranges from 0-30, sedation factor ranges from 0-30)
Safety and tolerability of CBD | Approximately 5 weeks
  Measured through monitoring adverse effects during the study, measured by number of adverse effects and severity of adverse effect.
Differences in alcohol consumption (measured by the Timeline Follow Back method) outside of the lab during treatment with CBD vs. placebo | 10 days
  Number of drinks, drinking days and binge drinking (≥ 4 drinks during a single day for females, ≥ 5 drinks during a single day for males)
Differences in alcohol craving (measured by Penn Alcohol Craving Scale) outside of the lab during treatment with CBD vs. placebo | 7 days
  Measures craving for alcohol (minimum score = 0; maximum score = 30; higher score indicates greater levels of craving)
Differences in self-reported anxiety (measured by modified Generalized Anxiety Disorder-7) outside of the lab during treatment with CBD vs. placebo | 7 days
  Measures generalized anxiety (Minimum score = 0; maximum score = 21; higher scores indicate higher levels of anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sloan, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada